CLINICAL TRIAL: NCT01327664
Title: A Multicenter, Open-label Study to Evaluate the Long Term Clinical Use of Treatment With AIN457 in Patients Completing Clinical Trials Investigating AIN457 for the Treatment of Non-infectious Intermediate, Posterior or Panuveitis
Brief Title: Study to Evaluate the Long Term Use of Treatment With AIN457 for Uveitis
Acronym: SUPPORT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study will not be initiated as planned.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals Corporation
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457C2399; 2010-021239-15 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-04-01 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Uveitis
Keywords: Quiescent uveitis; intermediate uveitis; panuveitis; posterior uveitis; uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Panuveitis; Uveitis, Posterior | interventions — secukinumab

ARMS (1):
- AIN457 300mg s.c every 2 weeks (Experimental)
  Interventions: Biological: AIN457

INTERVENTIONS:
Biological: AIN457

SUMMARY:
This study will provide patients who have completed the AIN457 Phase II and Phase III clinical trials in non-infectious uveitis continued access to treatment with AIN457 while collecting safety data and information on long term clinical use of treatment with AIN457.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand and communicate with the investigator and comply with the requirements for the study and must give a written, signed, and dated informed consent before any study assessment is performed
* Patient is currently enrolled in CAIN457A2208 or has completed the core and extension study treatment periods in the ongoing AIN457 phase III clinical trial Studies (e.g., CAIN457C2301 and CAIN457C2301E1)
* Willingness to discontinue AIN457 or be weaned from standard of care immunosuppressive therapy if recommended by the study investigator

Exclusion Criteria:

* Need for treatment with ocular procedures or systemic medications prohibited in this study including an alkylating agent or another biologic therapy other than AIN457
* Pregnant or nursing (lactating) women
* Women of childbearing potential unwilling to use protocol defined acceptable methods of contraception throughout the study and for 16 weeks after study drug discontinuation

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Participants with adverse events as a measure of safety and tolerability | up to 36 months
Proportion of patients achieving the criteria for clinically inactive posterior segment uveitis | up to 36 months
Mean time to achieve the criteria for clinically inactive posterior segment uveitis | up to 36 months

SECONDARY OUTCOMES:
Proportion of patients experiencing clinically active posterior segment uveitis in patients discontinuing AIN457 treatment | up to 36 months
Time to recurrence of clinically active posterior segment uveitis after discontinuation of AIN457 treatment | up to 36 months
Time to resolution of a recurrence of clinically active posterior segment uveitis in patients discontinuing AIN457 and treated only with the reinitiation of AIN457 | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals